CLINICAL TRIAL: NCT05213325
Title: Evaluation of Serum Interleukin 6 and 8 in Children With Acute Gastroentritis
Brief Title: Evaluation of Serum Interleukin 6 and 8 in Children With Acute Gastroenteritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, John Samuel Shaker, resident doctor at pediateric department sohag university hospital, Sohag University
Other Study IDs: Soh-Med-21-12-07
Record Dates: First submitted 2021-12-26; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Acute Gastroenteritis; Acute Diarrhea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Children with acute diarrhea
  Interventions: Diagnostic Test: Evaluation of serum levels of IL-6 and IL-8
- Control: Healthy control children
  Interventions: Diagnostic Test: Evaluation of serum levels of IL-6 and IL-8

INTERVENTIONS:
Diagnostic Test: Evaluation of serum levels of IL-6 and IL-8 — Evaluation of serum levels of IL-6 and IL-8 by Luminex Assay (multiplexed ELISA kits)

SUMMARY:
Cytokines, such as IL-6 and IL-8 can be used as markers of acute infections, including acute gastroenteritis. This study aims to evaluate serum levels of interleukins 6 and 8 in children with acute gastroenteritis.

ELIGIBILITY:
Group 1: Cases (Children with acute diarrhea)

Inclusion Criteria:

* Children aged 6 months to 5 years.
* Acute diarrhea: defined according to WHO criteria as the "passage of loose or watery stools at least three times in a 24 h period", lasts less than 14 days, with or without fever or vomiting, but considering the importance of change in stool consistency rather than frequency, and the usefulness of parental insight in deciding whether children have diarrhea or not.

Exclusion Criteria:

* Malnutrition or obesity
* History of antibiotic therapy in the last 72 hours.
* Acute diarrhea in association with systemic infections
* Malignancy
* Chronic diarrhea
* Autoimmune and autoinflammatory diseases.
* Chronic renal/liver failure
* Diabetes mellitus

Group 2: Controls (Healthy control children)

Inclusion Criteria:

• Healthy children aged 6 months to 5 years.

Exclusion Criteria:

* Acute diarrhea
* Malnutrition or obesity
* History of antibiotic therapy in the last 72 hours.
* Acute diarrhea in association with systemic infections
* Malignancy
* Chronic diarrhea
* Autoimmune and autoinflammatory diseases.
* Chronic renal/liver failure
* Diabetes mellitus

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children presented to the Pediatric Department and Outpatient Clinic at Sohag University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Serum level of Interleukin 6 | Within the first 3 days of acute diarrhea
  Difference in serum level of interleukin 6 between cases and control groups
Serum level of Interleukin 8 | Within the first 3 days of acute diarrhea
  Difference in serum level of interleukin 8 between cases and control groups

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muhsen K, Kassem E, Rubenstein U, Goren S, Ephros M, Shulman LM, Cohen D. No evidence of an increase in the incidence of norovirus gastroenteritis hospitalizations in young children after the introduction of universal rotavirus immunization in Israel. Hum Vaccin Immunother. 2019;15(6):1284-1293. doi: 10.1080/21645515.2019.1599522. Epub 2019 May 3. PMID 30945960
- [Background] Chen SM, Lin CP, Tsai JD, Chao YH, Sheu JN. The significance of serum and fecal levels of interleukin-6 and interleukin-8 in hospitalized children with acute rotavirus and norovirus gastroenteritis. Pediatr Neonatol. 2014 Apr;55(2):120-6. doi: 10.1016/j.pedneo.2013.05.008. Epub 2013 Jul 27. PMID 23899552
- [Background] Hamiel U, Bahat H, Kozer E, Hamiel Y, Ziv-Baran T, Goldman M. Diagnostic markers of acute infections in infants aged 1 week to 3 months: a retrospective cohort study. BMJ Open. 2018 Jan 24;8(1):e018092. doi: 10.1136/bmjopen-2017-018092. PMID 29371270